CLINICAL TRIAL: NCT01474915
Title: Aprepitant Versus Ondansetron in Preoperative Triple-therapy Treatment of Nausea and Vomiting
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sergio Bergese (Other)
Responsible Party: Sponsor-Investigator, Sergio Bergese, Associate Professor, Ohio State University
Organization: Ohio State University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2007H0053
Record Dates: First submitted 2011-11-08; First posted 2011-11-18 (Estimated); Results first posted 2013-12-03 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Postoperative Nausea and Vomiting (PONV); Nausea
Keywords: Neurosurgery
MeSH Terms: conditions — Postoperative Nausea and Vomiting; Nausea | interventions — Aprepitant; Ondansetron; Promethazine; Diphenhydramine; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Aprepitant (Active Comparator): Aprepitant is given orally, along with an oral or PO placebo depending on their group assignment for uniformity. Each patient will receive three drugs in their respective triple prophylactic medication plus an IV or oral placebo prior to induction of anesthesia.
  Triple therapy 40mg Aprepitant PO + IV placebo, 25mg Promethazine IV and 10mg dexamethasone IV
  Interventions: Drug: Aprepitant; Drug: Promethazine; Drug: Dexamethasone
- Ondansetron (Active Comparator): Ondansetron is given via IV, along with an oral or IV placebo depending on their group assignment for uniformity. Each patient will receive three drugs in their respective triple prophylactic medication (25mg promethazine, 10mg dexamethasone, and either 4mg ondansetron or 40mg aprepitant) plus an IV or oral placebo prior to induction of anesthesia.
  Triple therapy
  4mg Ondansetron IV + PO placebo, 25mg Promethazine IV and 10mg dexamethasone IV
  Interventions: Drug: Ondansetron; Drug: Promethazine; Drug: Dexamethasone

INTERVENTIONS:
Drug: Aprepitant — Subject will receive 40 mg of Aprepitant versus placebo PO before anesthesia induction
  Other Names: Emend
  Arms: Aprepitant
Drug: Ondansetron — Subject will receive 4 mg of Ondansetron IV versus placebo around anesthesia induction
  Other Names: Zofran
  Arms: Ondansetron
Drug: Promethazine — Subject will receive 25 mg of Promethazine IV around anesthesia induction
  Other Names: •Pentazine; •Phenadoz; •Phenergan; •Phenergan Fortis; •Promacot; •Promethegan
Drug: Dexamethasone — Subject will receive 10 mg of Dexamethasone IV around anesthesia induction
  Other Names: Decadron; Dexpak

SUMMARY:
This study is being done to determine the efficacies of two preventative drug combinations for postoperative nausea and vomiting in patients undergoing neurosurgery. The aim of this study is to compare the efficacy of using aprepitant instead of ondansetron in combination with dexamethasone and promethazine for post-operative nausea and vomiting prophylaxis. By completing this comparison study investigators will determine the most efficacious drug combination which will allow us to enhance the overall comfort and satisfaction of neurosurgical patients in the immediate postoperative period.

DETAILED DESCRIPTION:
One hundred-seventy-six (200) consecutive patients meeting the inclusion and exclusion criteria and who give written informed consent to participate in the study will be randomly assigned to one of two experimental groups using a 1:1 ratio. Patients in Group I will receive 25mg promethazine given intravenously (IV), 10mg dexamethasone given IV, 4mg ondansetron given intravenously, and a placebo pill given orally. Patients in Group II will receive 25mg promethazine given IV, 10mg dexamethasone given IV, 40mg aprepitant given orally, and an intravenous placebo. Thus all patients receive 25mg promethazine and 10mg dexamethasone. Group I will additionally receive 4mg ondansetron plus placebo PO and Group II will additionally receive 40mg aprepitant plus IV placebo. Because this is a double-blind study and because ondansetron is given intravenously whereas aprepitant is given orally, it is necessary to give patients an oral or IV placebo, depending on their group assignment for uniformity. Thus each patient will receive the three drugs in the PONV prophylactic triple cocktail, plus an IV or oral placebo prior to induction of anesthesia. See table below.

The following demographic and preoperative data about each patient in the two groups will be recorded:

Demographic and Preoperative Data Gender Systolic blood pressure, diastolic blood pressure, median blood pressure Age Smoking history PONV History Motion sickness history Surgery Anesthesia modality CPP Race ECG recording Hepatic function Renal function Past reactions to the study drugs

The duration of each surgery (anesthesia time) will be recorded for each patient. Patients will be continuously monitored in the post anesthesia care unit (PACU), surgical intensive care unit (SICU) and the medical floor for a total of 120 hours post operatively. Episodes of nausea, vomiting and administration of rescue therapy for either nausea or vomiting will be recorded and time stamped. In addition, the severity of the nausea or vomiting will be recorded. Nausea will be evaluated by the patient utilizing a standard verbal response scale (VRS) ranging from 0-10, 0 being no nausea and 10 being severe nausea. Vomiting will be evaluated by the investigator or nursing staff numerically as either 0, no vomiting, 1, mild vomiting, 2, moderate vomiting, or 3, severe vomiting. Rescue therapy for PONV episodes will consist of 4mg ondansetron. After the first 24hrs of starting the triple therapy antiemetic, ECG will be recorded as well as blood drawn for analysis.

Variables Primary Efficacy Variable The percentage of patients with no vomiting over 0-72 hours post operatively across the two treatment groups.

Secondary Efficacy Variables: Proportion of patients with a complete response during delayed (24-120 hours; days 2-5) and overall (0-120 hours; days 1-5) after neurological surgery and general anesthesia.

Proportion of patients with complete control, defined as no emetic episode, no need for rescue medication and no more than mild nausea overall (0-120 hours; days 1-5) after neurological surgery and general anesthesia.

Assess the severity of nausea and vomiting during acute (0-24 hours), delayed (24-120 hours) and overall (0-120 hours) intervals after neurological surgery and general anesthesia.

Assess the time to treatment failure (defined as time to first emetic episode and/or to first use of rescue medication).

Assess the time to first emetic episode.

Assess the time to significant nausea (defined as nausea rated ≥ 4 on a 0 to 10 verbal response scale or nausea that required rescue therapy).

Adverse Reactions to Treatment The incidence of any adverse reaction to treatment in the our two experimental groups will be recorded. In the ondansetron-treated patients (Group I), all cardiovascular, gastrointestinal, hepatic, integumentary and neurologic postoperative adverse events will be recorded and analyzed for cause. For instance, treatment-related diarrhea, headaches, fever, akathisia and acute dystonic reactions will be recorded and analyzed. Similarly, in the aprepitant-patients (Group II) all adverse events related to the digestive, hemic, lymphatic, nervous, cardiovascular and respiratory systems will be recorded and analyzed for cause.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* 18 to 85 years of age
* Scheduled for neurosurgery requiring opening of the cranium and dura at Ohio State University Medical Center and who consent in writing to participate in this study are eligible.

Exclusion Criteria:

* Patients will be excluded from this study if they are

  1. prisoners
  2. pregnant women
  3. mentally ill
  4. under the age of 18 or over the age of 85
  5. American Society of Anesthesiologist (ASA) classification V
  6. alcohol or drug abusers
  7. have a cerebral perfusion pressure (CPP) greater than 150 mmHg or less than 50 mmHg.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2007-06; Primary Completion 2012-12 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergio D Bergese, M.D., Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted at The Ohio State University Wexner Medical Center. It started in January of 2009 and ended in April of 2012.
Pre-assignment Details: Whenever a participant was enrolled into the study but later did not meet all the inclusion/exclusion criteria, they were excluded from the trial before assignment to groups.
Groups:
- Aprepitant: Aprepitant is given orally, along with an oral or PO placebo depending on their group assignment for uniformity. Each patient will receive three drugs in their respective triple prophylactic medication plus an IV or oral placebo prior to induction of anesthesia.
  Triple therapy 40mg Aprepitant PO + IV placebo, 25mg Promethazine IV and 10mg dexamethasone IV
  Aprepitant : Subject will receive 40 mg of Aprepitant versus placebo PO before anesthesia induction
  Dexamethasone : Subject will receive 10 mg of Dexamethasone IV around anesthesia induction
  Promethazine : Subject will receive 25 mg of Promethazine IV around anesthesia induction
- Ondansetron: Ondansetron is given via IV, along with an oral or IV placebo depending on their group assignment for uniformity. Each patient will receive three drugs in their respective triple prophylactic medication (25mg promethazine, 10mg dexamethasone, and either 4mg ondansetron or 40mg aprepitant) plus an IV or oral placebo prior to induction of anesthesia.
  Triple therapy
  4mg Ondansetron IV + PO placebo, 25mg Promethazine IV and 10mg dexamethasone IV
  Dexamethasone : Subject will receive 10 mg of Dexamethasone IV around anesthesia induction
  Ondansetron : Subject will receive 4 mg of Ondansetron IV versus placebo around anesthesia induction
  Promethazine : Subject will receive 25 mg of Promethazine IV around anesthesia induction
Period: Overall Study
Arm/Group | Aprepitant | Ondansetron
Started | 60 | 61
Completed | 50 | 51
Not Completed | 10 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aprepitant | Ondansetron | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 45 | 47 | 92
  >=65 years | 15 | 14 | 29
Age Continuous [Mean (Standard Deviation); unit: years] | 51.8136 (14.7) | 50.15 (16.4) | 50.9748 (15.6062)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 28 | 62
  Male | 26 | 33 | 59
Region of Enrollment [Number; unit: participants]
  United States | 60 | 61 | 121

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With a Complete Response/Complete Control During the First 24 Hours After Neurological Surgery Under General Anesthesia
Description: To assess the efficacy of triple therapy with Scopolamine, Ondansetron and Dexamethasone for prevention of post operative nausea and vomiting (PONV) in high risk patients during the first 24 hours after neurological surgery under general anesthesia.
  - Proportion of patients with a complete response/complete control during the first 24 hours after neurological surgery under general anesthesia.
  Complete Control is defined as no emetic episode, no need for rescue medication and no more than mild nausea overall after neurological surgery and general anesthesia.
  Complete Response is defined as no vomiting and no rescue therapy after neurological surgery and general anesthesia.
Time Frame: 24 hours post operatively
Population: Number of patients with Complete Control
Measure: Number; unit: participants
Groups:
- Aprepitant: Aprepitant is given orally (PO), along with an oral or PO placebo depending on their group assignment for uniformity. Each patient receives three drugs in their respective triple prophylactic medication plus an intravenous (IV) or oral placebo prior to induction of anesthesia.
  Triple therapy 40mg Aprepitant PO + IV placebo, 25mg Promethazine IV and 10mg dexamethasone IV
  Aprepitant : Subject receives 40 mg of Aprepitant versus placebo PO before anesthesia induction
  Dexamethasone : Subject receives 10 mg of Dexamethasone IV around anesthesia induction
  Promethazine : Subject receives 25 mg of Promethazine IV around anesthesia induction
- Ondansetron: Ondansetron is given via intravenous (IV), along with an oral (PO) or IV placebo depending on their group assignment for uniformity. Each patient receives three drugs in their respective triple prophylactic medication (25mg promethazine, 10mg dexamethasone, and either 4mg ondansetron or 40mg aprepitant) plus an IV or oral placebo prior to induction of anesthesia.
  Triple therapy
  4mg Ondansetron IV + PO placebo, 25mg Promethazine IV and 10mg dexamethasone IV
  Dexamethasone : Subject receives 10 mg of Dexamethasone IV around anesthesia induction
  Ondansetron : Subject receives 4 mg of Ondansetron IV versus placebo around anesthesia induction
  Promethazine : Subject receives 25 mg of Promethazine IV around anesthesia induction
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 50 | 51
participants
  Complete Control | 38 | 41
  Complete Response | 30 | 30

2. Secondary Outcome: Post Operative Nausea and Vomiting (PONV) Scores on a Verbal Response Scale
Description: To assess the efficacy of triple therapy with Scopolamine, Ondansetron and Dexamethasone for prevention of post operative nausea and vomiting (PONV) in high risk patients during a delayed period after neurological surgery under general anesthesia.
  - Assess the severity of nausea and vomiting during the first 24 hours after neurological surgery.
  Nausea is evaluated by a standard verbal response scale (VRS) ranging from 0-10, 0 being no nausea and 10 being severe nausea. Vomiting is evaluated by the investigator or nursing staff numerically as either 0, no vomiting;, 1, mild vomiting;, 2, moderate vomiting;, or 3, severe vomiting.
Time Frame: 24 hours post-operatively
Population: Severity of nausea and vomiting
Measure: Mean (Full Range); unit: units on a scale
Groups:
- Aprepitant: Aprepitant is given orally (PO), along with an oral or PO placebo depending on their group assignment for uniformity. Each patient will receive three drugs in their respective triple prophylactic medication plus an intravenous (IV) or oral placebo prior to induction of anesthesia.
  Triple therapy 40mg Aprepitant PO + IV placebo, 25mg Promethazine IV and 10mg dexamethasone IV
  Aprepitant : Subject receives 40 mg of Aprepitant versus placebo PO before anesthesia induction
  Dexamethasone : Subject receives 10 mg of Dexamethasone IV around anesthesia induction
  Promethazine : Subject receives 25 mg of Promethazine IV around anesthesia induction
Arm/Group | Aprepitant | Ondansetron
Number analyzed (Participants) | 50 | 51
units on a scale
  Nausea episodes | 1 [1 to 2] | 1 [1 to 2]
  Vomiting episodes | 1.5 [1 to 2] | 1.5 [1 to 3]

ADVERSE EVENTS:
Arm/Group | Aprepitant | Ondansetron
Serious Adverse Events (participants affected / at risk) | 2/60 | 3/61
Other Adverse Events (participants affected / at risk) | 0/60 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aprepitant (N=60) | Ondansetron (N=61)
Fever (General disorders) | 0 (0) | 1 (1) — Unrelated fever resulting in re-hospitalization
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) — Unrelated deep vein thrombosis resulting in prolonged hospitalization
Cerebrovascular Hematoma (Nervous system disorders) | 2 (2) | 0 (0) — Unrelated cerebrovascular hematoma resulting in additional surgical procedure for evacuation
Cerebrospinal fluid leak (Nervous system disorders) | 0 (0) | 1 (1) — Unrelated cerebrospinal fluid leak resulting in additional procedure

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No